CLINICAL TRIAL: NCT02031042
Title: Sentinel Node Biopsy Before and/or After Neoadjuvant Chemotherapy in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Stockholm South General Hospital (Other)
Collaborators: Swedish Breast Cancer Group (Other)
Responsible Party: Principal Investigator, Linda Zetterlund, MD, PhD student, Stockholm South General Hospital
Other Study IDs: 2010/441-31/4
Record Dates: First submitted 2013-12-19; First posted 2014-01-09 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: neoadjuvant chemotherapy; breast cancer; sentinel lymph node biopsy; false negative rate; identification rate
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate if sentinel lymph node biopsy is a reliable staging tool for breast cancer patients planned for neoadjuvant chemotherapy (=before breast surgery) and if, in that case, it is safe to omit axillary lymph node dissection if the sentinel lymph node is free of metastasis.

DETAILED DESCRIPTION:
Sentinel lymph node biopsy (SLNB) was introduced in the late 1990´s and has become standard procedure for staging of the axilla in early stage breast cancer associated with significantly less arm morbidity than axillary lymph node dissection (ALND).

Neoadjuvant chemotherapy (NAC) given before breast surgery is indicated for locally advanced breast cancer but is increasingly used for early stage breast cancer with the purpose of downstaging the tumor and thereby possibly enabling breast conserving surgery. Traditionally, the standard axillary staging tool has been ALND although up to 50 per cent of the patients at diagnosis do not have any metastases in their axillary lymph nodes. In addition, NAC can eradicate metastases in the axillary lymph nodes in up to 40 per cent of the patients.

SLNB has therefore been evaluated in the neoadjuvant setting both before and after NAC but is still controversial and the timing debated.

This is a Swedish prospective multi-institutional study without any comparison goup. The comparison is between the findings in the SLNB and the following ALND performed after NAC in all patients.

If the patient is clinically node-negative at diagnosis a SLNB is performed before (without frozen section) and after NAC (substudy I). The reasons for repeating SLNB both before and after NAC are 1) to find out what happens during NAC 2) if it is possible to identify a repeat SLNB and 3) if it is reliable.

If the patient is node-positive at diagnosis (cytologically verified lymph node metastasis) SLNB is performed after NAC together with the breast operation and ALND (substudy II). When SLNB is performed after NAC, the sentinel lymph nodes are also analysed with frozen section in order to validate the method after chemotherapy. Both blue dye and radiolabelled isotope for localisation of the sentinel lymph node is recommended but lymphoscintigraphy is optional.

All consecutive clinically node-negative (or with unclear nodal status after ultrasound and cytology) patients planned for NAC will have oral and written information about the study by the responsible surgeon. After accepting to participate, the patient is asked to sign a written consent. Patients with a cytologically verified lymph node metastasis/es at diagnosis will be informed and asked to participate in substudy II after completion of NAC.

According to the statistical analysis, and with an expected loss of 10 per cent, a sample size of 220 patients is needed in substudy I to show that the false negative rate is less than 10 per cent. If we include 200 patients and 50 per cent are lymph node positive at diagnosis then the estimation of false negative rate will be based on 100 individuals. If we estimate the true false negative rate to be 8 per cent, then the precision with 80 per cent power will be +/- 7 per cent units (2-sided test with 95 per cent confidence interval).

The Central Contact (PI) is responsible for data collection, management and analysis. Each protocol will be sent together with a written consent and copies of all relevant histopathological reports to the PI, who will control for missing or incongruent data and if so, ask the responsible investigator on that institution/hospital to complement the missing data from the patients journal (copies of medical records or histopathological reports).

ELIGIBILITY:
Inclusion Criteria:

* clinically node-negative (or unclear nodal status) substudy I
* signed consent from the study participant

Exclusion Criteria:

* inflammatory breast cancer
* cytologically verified lymph node metastasis/es at diagnosis (substudy I), but these patients can be included in substudy II
* patients not able to give an informed consent
* hypersensitivity or allergy against blue dye or isotope

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically verified breast cancer planned for neoadjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2010-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
False negative rate | Up to two years
  The rate of patients with no metastasis/ses in their sentinel lymph node/s before neoadjuvant chemotherapy (NAC) but metastasis/ses in the nodes from the axillary lymph node dissection performed after NAC will be analysed. In substudy II we also investigate the false negative rate in sentinel lymph node biopsies performed after NAC if the patient had positive lymph nodes at diagnosis.

SECONDARY OUTCOMES:
Identification rate | Up to two years
  The number of successful sentinel lymph node biopsies among the total number of attempted biopsies. Will be analyses both before and after neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Linda H Zetterlund, PhD, Principal Investigator — Dep. of Medical Research and Education, Karolinska Institutet (KI), Stockholm, Sweden; Fuat Celebioglu, PhD, Study Chair — Dep. of Medical Research and Education, KI, Stockholm, Sweden; Jan Frisell, Professor, Study Chair — Dep. of Molecular Medicine and Surgery, KI, Stockholm, Sweden
Locations (20):
- Sweden (20):
  - Falu lasarett, Falun
  - Sahlgrenska Universitetssjukhuset, Sahlgrenska, Gothenburg
  - Länssjukhuset i Halmstad, Halmstad
  - Helsingborgs lasarett, Helsingborg
  - Blekingesjukhuset Karlskrona, Karlskrona
  - Centralsjukhuset i Karlstad, Karlstad
  - Centralsjukhuset i Kristianstad, Kristianstad
  - Universitetssjukhuset i Linköping, Linköping
  - Skånes Universitetssjukhus, Lund, Lund
  - Skånes Universitetssjukhus, Malmö, Malmo
  - Universitetssjukhuset i Örebro, Örebro
  - Capio St Görans Sjukhus, Stockholm
  - Södersjukhuset/Stockholm South General Hospital, Stockholm
  - Karolinska Universitetssjukhuset i Solna, Stockholm
  - Länssjukhuset Sundsvall-Härnösand, Sundsvall
  - NU-sjukvården, Uddevalla sjukhus, Uddevalla
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska sjukhuset i Uppsala, Uppsala
  - Centrallasaretttet i Växjö, Vaxjo
  - Centrallasarettet i Västerås, Västerås

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuerer HM, Sahin AA, Hunt KK, Newman LA, Breslin TM, Ames FC, Ross MI, Buzdar AU, Hortobagyi GN, Singletary SE. Incidence and impact of documented eradication of breast cancer axillary lymph node metastases before surgery in patients treated with neoadjuvant chemotherapy. Ann Surg. 1999 Jul;230(1):72-8. doi: 10.1097/00000658-199907000-00011. PMID 10400039
- [Background] Bear HD, Anderson S, Brown A, Smith R, Mamounas EP, Fisher B, Margolese R, Theoret H, Soran A, Wickerham DL, Wolmark N; National Surgical Adjuvant Breast and Bowel Project Protocol B-27. The effect on tumor response of adding sequential preoperative docetaxel to preoperative doxorubicin and cyclophosphamide: preliminary results from National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2003 Nov 15;21(22):4165-74. doi: 10.1200/JCO.2003.12.005. Epub 2003 Oct 14. PMID 14559892
- [Background] Mamounas EP, Brown A, Anderson S, Smith R, Julian T, Miller B, Bear HD, Caldwell CB, Walker AP, Mikkelson WM, Stauffer JS, Robidoux A, Theoret H, Soran A, Fisher B, Wickerham DL, Wolmark N. Sentinel node biopsy after neoadjuvant chemotherapy in breast cancer: results from National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2005 Apr 20;23(12):2694-702. doi: 10.1200/JCO.2005.05.188. PMID 15837984
- [Background] Xing Y, Foy M, Cox DD, Kuerer HM, Hunt KK, Cormier JN. Meta-analysis of sentinel lymph node biopsy after preoperative chemotherapy in patients with breast cancer. Br J Surg. 2006 May;93(5):539-46. doi: 10.1002/bjs.5209. PMID 16329089
- [Background] Schrenk P, Hochreiner G, Fridrik M, Wayand W. Sentinel node biopsy performed before preoperative chemotherapy for axillary lymph node staging in breast cancer. Breast J. 2003 Jul-Aug;9(4):282-7. doi: 10.1046/j.1524-4741.2003.09406.x. PMID 12846861
- [Background] Papa MZ, Zippel D, Kaufman B, Shimon-Paluch S, Yosepovich A, Oberman B, Sadetzki S. Timing of sentinel lymph node biopsy in patients receiving neoadjuvant chemotherapy for breast cancer. J Surg Oncol. 2008 Nov 1;98(6):403-6. doi: 10.1002/jso.21128. PMID 18683193
- [Background] Kuehn T, Bauerfeind I, Fehm T, Fleige B, Hausschild M, Helms G, Lebeau A, Liedtke C, von Minckwitz G, Nekljudova V, Schmatloch S, Schrenk P, Staebler A, Untch M. Sentinel-lymph-node biopsy in patients with breast cancer before and after neoadjuvant chemotherapy (SENTINA): a prospective, multicentre cohort study. Lancet Oncol. 2013 Jun;14(7):609-18. doi: 10.1016/S1470-2045(13)70166-9. Epub 2013 May 15. PMID 23683750
- [Background] Boughey JC, Suman VJ, Mittendorf EA, Ahrendt GM, Wilke LG, Taback B, Leitch AM, Kuerer HM, Bowling M, Flippo-Morton TS, Byrd DR, Ollila DW, Julian TB, McLaughlin SA, McCall L, Symmans WF, Le-Petross HT, Haffty BG, Buchholz TA, Nelson H, Hunt KK; Alliance for Clinical Trials in Oncology. Sentinel lymph node surgery after neoadjuvant chemotherapy in patients with node-positive breast cancer: the ACOSOG Z1071 (Alliance) clinical trial. JAMA. 2013 Oct 9;310(14):1455-61. doi: 10.1001/jama.2013.278932. PMID 24101169
- [Derived] Zetterlund L, Celebioglu F, Axelsson R, de Boniface J, Frisell J. Swedish prospective multicenter trial on the accuracy and clinical relevance of sentinel lymph node biopsy before neoadjuvant systemic therapy in breast cancer. Breast Cancer Res Treat. 2017 May;163(1):93-101. doi: 10.1007/s10549-017-4163-2. Epub 2017 Feb 17. PMID 28213781
- See also: Homepage for the Swedish Breast Surgical Association — http://sffb.se